CLINICAL TRIAL: NCT04763928
Title: A Phase 2, Prospective, Multi-center Intervention Trial in Patients With Acute Myeloid Leukemia Secondary to Myeloproliferative Neoplasms Unfit for Intensive Chemotherapy Investigating a Treatment Combination Including Decitabine and Venetoclax
Brief Title: Trial in AML Secondary to MPNs Patients, Unfit for Intensive Chemotherapy, Investigating a Treatment Combination Including Decitabine and Venetoclax
Acronym: ENABLE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML2420
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VenDec (Experimental): Patients will receive a combination of VENETOCLAX (400 mg per day orally on days 1 to 28 of 28-days courses) and DECITABINE (20 mg/sqm intravenously on days 1 to 5 of 28-days courses)
  Interventions: Drug: Venetoclax+Decitabine

INTERVENTIONS:
Drug: Venetoclax+Decitabine — Patients will receive treatment with a combination of decitabine and venetoclax as follows:
  * Decitabine 20 mg/sqm intravenously on days 1 to 5 of 28-days courses
  * Venetoclax 400 mg per day orally on days 1 to 28 of 28-days courses; a dose escalation period is provided at first cycle (ramp-up) in which VEN is administered as follows: 100 mg on day -2, 200 mg on day -1, and 400 mg on day 1, a dose that is continued subsequently, daily, for 28-day cycles.
  In case of achievement of response, the treatment will be continued until disease progression or death by other causes.

SUMMARY:
Prospective, multi-center, intervention, open clinical trial for the treatment of AML secondary to MPN in patients unfit for intensive chemotherapy investigating a combination regimen including VEN and DEC.

DETAILED DESCRIPTION:
Prospective, multi-center, intervention, open clinical trial for the treatment of AML secondary to MPN in patients unfit for intensive chemotherapy, investigating a combination regimen including VEN and DEC to improve the survival outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AML secondary to myeloproliferative neoplasms (sAML), untreated, newly diagnosed, according to WHO 2016 criteria based on conventional cytological, cytogenetic, and immunophenotypic disease characterization
2. Patients unfit for intensive treatment modalities at the discretion of the investigator.
3. ECOG performance status 0-2 or disease-related reversible ECOG 3 score following adequate supportive care.
4. Signed written informed consent according to ICH/EU/GCP and national local laws.
5. Males enrolled in the study with partners who are women of childbearing potential, must be willing to use an acceptable barrier contraceptive method during the trial

Exclusion Criteria:

1. Diagnosis of de novo AML
2. Pre-existing, uncontrolled pathology such as heart failure (congestive/ischaemic, acute myocardial infarction within the post 3 months, untreatable arrhythmias, NYHA classes III and IV), sever liver disease with total bilirubin ≥2,5 x ULN and/or ALT>3 ULN (unless attributable to AML), acute or chronic pancreatitis, kidney function impairment with Creatinine Clearance (CrCl) level <30ml/min (calculated by Cockcroft Gault formula) (unless attributable to AML) and severe neuropsychiatric disorder that impairs the patient's ability to understand and sign the informed consent or to cope with the intended treatment plan. For altered liver, pancreas and kidney function tests, eligibility criteria can be reassessed at 24-96 hours, following adequate supportive measures.
3. Pre-existing HIV positive serology (i.e. already known before enrolment). The participation to the study will require serology testing for HIV positivity at baseline: in case of HIV positivity or refusal to perform HIV testing, the patient will be considered not eligible.
4. Uncontrolled bacterial or fungal infections
5. QTc >470 msec on screening ECG (Fridericia's formula)
6. A history of cancer that is not in remission phase following surgery and/or chemotherapy and/or radiotherapy with life expectancy < 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy of VEN-DEC regimen (event free survival) | at 1 year
  Evaluation of the event free survival at 1 year of an experimental VEN-DEC combination arm in patients with AML secondary to MPN and unfit for intensive therapeutic strategy

CONTACTS AND LOCATIONS:
Locations (33):
- Italy (33):
  - Ematologia A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ematologia AOU delle Marche, Ancona
  - Ematologia AOU Policlinico Bari, Bari
  - Ematologia ASST Papa Giovanni XXIII, Bergamo
  - Ematologia IRCCS AOU di Bologna, Bologna
  - Ematologia ASST Spedali Civili di Brescia, Brescia
  - Ematologia Businco, Cagliari
  - Ematologia Istituto Oncologico Veneto IRCCS, Castelfranco Veneto
  - Ematologia AOU Policlinico Rodolico-San Marco, Catania
  - Ematologia A.O.U Arcispedale S.Anna, Cona
  - Ematologia Ospedale A.Carle, Cuneo
  - Az. Ospedaliero - Universitaria Careggi, Florence
  - Ematologia IRCCS Ospedale Policlinico San Martino, Genova
  - Ematologia AOU di Modena, Modena
  - Ematologia AORN Cardarelli, Napoli
  - Ematologia Federico II, Napoli
  - Ematologia P.O. A.Tortora, Pagani
  - Ematologia AOU Policlinico Giaccone, Palermo
  - Ematologia Santa Maria della Misericordia, Perugia
  - Ematologia PO Santo Spirito ASL Pescara, Pescara
  - Ematologia Ospedale S.M.delle Croci, Ravenna
  - Ematologia AOU S.Andrea, Roma
  - Ematologia Fondazione PTV, Roma
  - Ematologia Ospedale Sant'Eugenio, Roma
  - Ematologia Policlinico Gemelli, Roma
  - Ematologia Policlinico Umberto I, Roma
  - Ematologia Policlinico Santa Maria alle Scotte, Siena
  - Ematologia A.O.S. Maria Di Terni, Terni
  - Ematologia Città della Salute e della Scienza, Torino
  - Ematologia ORDINE MAURIZIANO DI TORINO, Torino
  - Ematologia Santa Maria della Misericordia, Udine
  - Ematologia ASST SETTE LAGHI, Varese
  - Ematologia Ospedale Belcolle, Viterbo